CLINICAL TRIAL: NCT00842101
Title: Effect of Reamed Intramedullary Nails in Tibial Fractures as a Factor of Rising Intracompartmental Pressures: A Clinical Study
Brief Title: Compartmental Overpressures Associated to Reamed Intramedullary Nails
Status: Completed | Type: Observational
Sponsor: University of Andorra (Other)
Responsible Party: JOSE IGNACIO TORRERO, ORTHOPAEDIC AND TRAUMA UNIT. ANDORRA´S HOSPITAL
Other Study IDs: UA002
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Tibial Fractures
Keywords: Intramedullary nails; Compartmental syndrome; Fractures
MeSH Terms: conditions — Tibial Fractures; Compartment Syndromes; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pressure monitor: Tibial Fracture
  Interventions: Device: Quick Pressure Monitor

INTERVENTIONS:
Device: Quick Pressure Monitor — The monitor measures actively the actual pressure inside the compartment affected.
  Other Names: Slit catheter

SUMMARY:
The purpose of this study is to determine the effect of reamed intramedullary nails in tibial shaft fractures (as a standard treatment), in raising intracompartmental pressures and therefore determine if they are a risk factor for compartmental syndrome.

DETAILED DESCRIPTION:
Compartmental overpressure is a serious problem in relation to the treatment of tibial shaft fractures. When reamed intramedullary nails are used, the risk of suffering a compartmental syndrome must be in mind of surgeons. Diagnostic of compartmental syndrome could be difficult just after the surgical intervention, because the patient is under conditions of regional anesthesia or opioids and analgesics, which could mask the symptomatology. In fact, when there is a great suspicion of this syndrome, we recommend measuring compartmental pressures; therefore, physicians might apply the term delta-P value, which is the result of the mean arterial pressure minus compartmental pressure. If this one is less than 30 mm Hg, a fasciotomy should be performed even when the clinical diagnostic is not clear.

ELIGIBILITY:
Inclusion Criteria:

* Tibial shaft fractures treated with intramedullary reamed nails

Exclusion Criteria:

* Tibial fractures treated with other types of fixation or nails not reamed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with tibial shaft fractures
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-12; Primary Completion 2008-04 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
intracompartmental pressures | 0-2 hours

CONTACTS AND LOCATIONS:
Overall Officials: JOSE I TORRERO, M.D., Principal Investigator — Orthopaedic and Trauma Unit. Andorra´s Hospital
Locations (1):
- Orthopaedic and Trauma Unit. Nostra Senyora de Meritxell Hospital, Les Escaldes, Andorra